CLINICAL TRIAL: NCT00348595
Title: Phase I/II Double Blinded Randomized Study to Determine the Tolerability and Efficacy of 2 Different Doses of Revlimid (CC-5013, Lenalidomide) in Biochemically Relapsed Prostate Cancer Patients (M0) After Local Treatment
Brief Title: Study of 2 Different Doses of Revlimid in Biochemically Relapse Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: J0798; RV-PCA-PI-069; NA_00013597 (Other: JHM IRB); J0798 (Other: JHM IRB)
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Results first posted 2019-04-12 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 5mg/day Arm: one 5 mg active Revlimid capsule and one 25 mg matched placebo capsules PO QAM (every morning) (at approximately the same time) days 1-21 days (28-day cycles).
  Interventions: Drug: Revlimid
- 2 (Active Comparator): 25 mg/day Arm: one 25 mg active Revlimid capsule and one 5 mg matched placebo capsule PO QAM (every morning) (at approximately the same time) days 1-21 (28 day cycles).
  Interventions: Drug: Revlimid

INTERVENTIONS:
Drug: Revlimid — one 5 mg/day capsule or one 25 mg/day capsule with matched placebo capsule day 1-21 (28 day cycle)
  Other Names: Lenalidomide

SUMMARY:
The primary objectives of the study are:

* To evaluate feasibility, safety and tolerance of 6 months administration of Revlimid at 5mg/day and 25mg/day, given orally in subjects with prostate cancer with evidence of biochemical relapse (M0) following local treatment (i.e., surgery or radiation).
* To assess the rate of PSA (prostatic specific antigen) progression at 6 months after treatment with 5mg/day and 25mg/day of Revlimid (CC-5013) in patients with evidence of biochemical relapse after local therapy.

The secondary objectives of the study are:

* To provide preliminary assessments on the effects of Revlimid (CC-5013) at 5mg/day and 25mg/day on various PSA constructs in the subject population (i.e., PSADT [Prostatic Specific Antigen Doubling Time] and PSA slope) by comparing pre and post treatment patterns in each arm.
* To evaluate preliminary pharmacodynamic correlations between serum revlimid concentrations and toxicity, PSA constructs and other evidence of disease progression.

DETAILED DESCRIPTION:
Carcinoma of the prostate in the most commonly diagnosed malignancy among men in this country with approximately 232,090 new cases expected to be diagnosed in 2005. Unfortunately, despite local treatment, many men will demonstrate evidence of PSA recurrence. At the present time, there is no standard treatment fo these patients. The management of patients with PSA recurrence remains greatly controversial. Androgen deprivation is frequently employed in patients with evidence of rising PSA levels despite the fact that the effects on quantity and quality of life of androgen deprivation therapy at this stage, remains un-established. Toxicity of androgen deprivation therapy is a major factor to be considered in the decision process of employing the modality of treatment in patients with no symptoms associated with this disease. Because patients with biochemical relapse are mostly asymptomatic and typically have long survivals and disease free survivals, mush of the focus of new drug development has been with the use of non-cytotoxic compounds. This study is intended to provide preliminary evidence of a biological effect in a dose response manner assessing the effects of Revlimid (CC-5013) on PSA.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of adenocarcinoma of the prostate (M0) with evidence of biochemical relapse after local therapy (i.e., surgery, radiation therapy, or both.) Baseline PSA must be greater or equal to 1 ng/ml.
* Confirmed rise in PSA shown by 2 PSA values at least 1 month apart, higher than a reference value noted within 6 months of study entry. Interim PSA values during the immediate pre-study six-month interval may demonstrate a "fluctuation" including a decline, however the study baseline PSA must have shown a rise within the pre-study 6-months period. Baseline PSA's must be determined within 4 weeks of study entry.
* All previous local modalities of treatment, including radiation and surgery, must have been discontinued at least 4 weeks prior to treatment in this study. May have received prior systemic chemotherapy, hormonal therapy, biologic or vaccine therapy. All treatment must have been discontinued for more than 6 months prior to study entry.
* Patients receiving intermittent hormonal therapy for their rising PSA state are considered eligible if testosterone level is above 150 ng/dl and treatment was discontinued greater than 6 months
* No clinical or radiological evidence of distant metastases (excluding prostascint scan).
* Serum testosterone > 150 ng/ml
* Disease free of prior malignancies for more than 5 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the breast.
* Able to take aspirin (ASA 81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use low molecular weight heparin). Lenalidomide increases the risk of thrombotic events in patients who are at high risk or with a history a thrombosis, in particular when combined with other drugs known to cause thrombosis.

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
* Known hypersensitivity to thalidomide.
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Any prior use of Revlimid® (CC-5013).
* Concurrent use of other anti-cancer agents or treatments.
* Known brain metastases.
* Known positive for HIV or infectious hepatitis, type A, B or C.
* Any evidence of metastatic disease.
* Any increase in PSA while receiving neo-adjuvant or adjuvant therapy or intermittent hormonal therapy.
* More than one prior biologic or vaccine therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2006-07-20 (Actual); Primary Completion 2016-06-29 (Actual); Study Completion 2016-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mario A Eisenberger, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- The Harry and Jeanette Weinberg Building, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 17 subjects were screen failures
Groups:
- Revlimid 5mg/Day: One 5 mg active Revlimid capsule and one 25 mg matched placebo capsule given by mouth daily in the morning (at approximately the same time) on days 1-21 (28-day cycles).
- Revlimid 25mg/Day: One 25 mg active Revlimid capsule and one 5 mg matched placebo capsule given by mouth daily in the morning (at approximately the same time) on days 1-21 (28-day cycles).
Period: Overall Study
Arm/Group | Revlimid 5mg/Day | Revlimid 25mg/Day
Started | 26 | 34
Completed | 21 | 26
Not Completed | 5 | 8
Not completed — Adverse Event | 5 | 8

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were only recorded for patients who entered the study.
Groups:
- Revlimid 5mg/Day: One 5 mg active Revlimid capsule and one 25 mg matched placebo capsule given by mouth daily in the morning (at approximately the same time) on days 1-21 (28-day cycles), repeated monthly for 6 months or until dose-limiting toxicity or disease progression, as defined in the protocol.
- Revlimid 25mg/Day: One 25 mg active Revlimid capsule and one 5 mg matched placebo capsule given by mouth daily in the morning (at approximately the same time) on days 1-21 (28-day cycles), repeated monthly for 6 months or until dose-limiting toxicity or disease progression, as defined in the protocol.
- Total: Total of all reporting groups
Arm/Group | Revlimid 5mg/Day | Revlimid 25mg/Day | Total
Number analyzed (Participants) | 26 | 34 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (7.1) | 63.1 (7.2) | 63.4 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 26 | 34 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 34 | 60
Gleason score [Mean (Standard Deviation); unit: units on a scale] — The Gleason score ranges from 2-10 with a higher score reflecting less-differentiated tumors with worse prognosis. The total score is a sum of two numbers which are based on the microscopic appearance of cells. The first number is the score based on the dominant, cell morphology (scored 1-5) and the second number is based on the highest grade of the non-dominant cell pattern (scored 1-5).
  units on a scale | 7.1 (1.0) | 7.3 (1.1) | 7.2 (1.05)
Local therapy [Count of Participants; unit: Participants]
  Radical prostatectomy | 12 | 12 | 24
  Radiation therapy | 4 | 8 | 12
  Surgery and Radiation therapy | 10 | 14 | 24
  Prior androgen deprivation therapy | 8 | 11 | 19
Serum testosterone [Mean (Full Range); unit: (ng/dL)] | 374 [148 to 564] | 342 [175 to 569] | 358 [148 to 569]
Prostate Specific Antigen (PSA) [Mean (Standard Deviation); unit: ng/mL] | 11.9 (11.9) | 12.4 (13.6) | 12.2 (12.8)
PSA doubling time (PSADT) [Count of Participants; unit: Participants]
  < 3 months | 6 | 10 | 16
  3-8.9 months | 13 | 16 | 29
  ≥ 9 months | 7 | 8 | 15
Pre-treatment PSA slopes [Mean (Full Range); unit: log PSA/month] | 0.16 [0.11 to 0.21] | 0.18 [0.13 to 0.23] | 0.17 [0.11 to 0.23]

OUTCOME MEASURES:

1. Primary Outcome: Safety, Feasibility and Tolerance of Revlimid as Assessed by Number of Participants Experiencing Grade 3 and 4 Adverse Events.
Description: Number of participants experiencing Grade 3 and 4 adverse events as defined by the National Cancer Institute Common Toxicity Criteria version 3.0
Time Frame: 6 months post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Revlimid 5mg/Day | Revlimid 25mg/Day
Number analyzed (Participants) | 26 | 34
Participants | 3 | 10

2. Primary Outcome: Number of Participants With Prostate-specific Antigen (PSA) Progression
Description: Number of participants with greater than or equal to 25% increase in PSA at 6 months
Time Frame: 6 months post-intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Revlimid 5mg/Day | Revlimid 25mg/Day
Number analyzed (Participants) | 26 | 34
Participants | 7 | 5

3. Primary Outcome: Change in of PSA Slope
Description: Mean change in PSA slope from baseline to 6 months. PSA slope was calculated using the regression of log PSA over 6 months in each patient. A negative mean change in PSA slope reflects a better outcome.
Time Frame: Change from baseline to 6 months post-intervention
Measure: Mean (95% Confidence Interval); unit: log PSA
Arm/Group | Revlimid 5mg/Day | Revlimid 25mg/Day
Number analyzed (Participants) | 26 | 34
log PSA | -0.033 [-0.11 to 0.04] | -0.172 [-0.24 to -0.11]

4. Secondary Outcome: Plasma Concentration of Revilimid at Steady State
Description: Mean plasma concentration (ng/mL) of Revilimid at steady state (Day 21 of second treatment cycle)
Time Frame: Day 21 of second treatment cycle
Population: Data was only evaluable in 20/26 and 27/34 participants from the 5mg and 25mg arms, respectively.
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Revlimid 5mg/Day | Revlimid 25mg/Day
Number analyzed (Participants) | 20 | 27
ng/mL | 12.67 [6.1 to 19.2] | 65.14 [24.3 to 106.0]

ADVERSE EVENTS:
Time Frame: Collected monthly, up to 44 months
Arm/Group | Revlimid 5mg/Day | Revlimid 25mg/Day
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/34
Serious Adverse Events (participants affected / at risk) | 3/26 | 10/34
Other Adverse Events (participants affected / at risk) | 26/26 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Revlimid 5mg/Day (N=26) | Revlimid 25mg/Day (N=34)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 5 (5)
venous thromboembolism (Vascular disorders) | 2 (2) | 2 (2)
Fatigue (Nervous system disorders) | 1 (1) | 1 (1)
Severe Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Revlimid 5mg/Day (N=26) | Revlimid 25mg/Day (N=34)
anemia (Blood and lymphatic system disorders) | 7 (7) | 10 (10)
Constipation (Gastrointestinal disorders) | 10 (10) | 15 (15)
Fatigue (Nervous system disorders) | 12 (12) | 29 (29)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (11) | 14 (14)
Increased of SGOT (Investigations) | 2 (2) | 8 (8)
Muscular Cramping (Nervous system disorders) | 5 (5) | 14 (14) — Leg and or Hand
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 8 (8)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 9 (9)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8) | 15 (15)
Rash (Skin and subcutaneous tissue disorders) | 7 (7) | 15 (15)
Thrombocytopenia (Blood and lymphatic system disorders) | 4/4 (4) | 8 (8)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 5 (5)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 5 (5)
Anal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 6 (6)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Blurred Vision (Eye disorders) | 1 (1) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 5 (5)
Dizziness (Nervous system disorders) | 4 (4) | 5 (5)
Dry Eye (Eye disorders) | 2 (2) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 5 (5)
Dry Skin (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5)
Flushing (Vascular disorders) | 0 (0) | 4 (4) — Facial Flushing
Headache (Nervous system disorders) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes